CLINICAL TRIAL: NCT06195176
Title: Randomized Clinical Trial: Effect of an Exercise Routine on Postoperative Shoulder Pain in Total Laparoscopic Hysterectomy
Brief Title: Randomized Clinical Trial: Effect of an Exercise Routine on Postoperative Shoulder Pain in Laparoscopic Hysterectomy
Acronym: ERPOSP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes (Other Government)
Responsible Party: Principal Investigator, Andrea Alicia Olguin Ortega, MD MSC, Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-1-40
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Pain; Laparoscopic Hysterectomy for Benign Conditions
Keywords: LAPAROSCOPIC HYSTERECTOMY; SHOULDER PAIN; EXERCISE; POSTOPERATIVE PAIN
MeSH Terms: conditions — Pain, Postoperative; Shoulder Pain; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHOULDER EXERCISES (Experimental): Patients randomized to the exercise routine group will be instructed, upon recovery, about the exercise routine. The routine consists of lifting the shoulders as high as possible towards the ears, holding for 3 seconds, and then resting. This should be repeated 10 times at the beginning of each hour during the immediate postoperative period while on the hospital ward. The routine will be suspended at night. The procedure will be standardized, as the principal investigators will personally explain and demonstrate it to all involved individuals who are responsible for explaining it to the patients. In-person reminders will be made, and pain in the shoulders, incisions, and abdomen will be recorded at 6 hours and 24 hours postoperatively, as well as during the follow-up consultations on day post-surgery
  Interventions: Other: Shoulder exercises
- HAND EXERCISES (Sham Comparator): Patients randomized to the exercise routine group will be instructed, upon recovery, about the exercise routine. The sham routine consists of tightly opening and closing the hands, holding for 3 seconds, and then resting. This should be repeated 10 times at the beginning of each hour during the immediate postoperative period while on the hospital ward. The routine will be suspended at night. The procedure will be standardized, as the principal investigator will personally explain and demonstrate it to all individuals responsible for instructing the patients. In-person reminders will be issued, and pain in the shoulders, incisions, and abdomen will be recorded at 6 hours and 24 hours postoperatively, as well as during the follow-up consultations on the 7th day after surgery.
  Interventions: Other: Hand exercises

INTERVENTIONS:
Other: Shoulder exercises — Operational Definition:
  * Lift the shoulders as high as possible toward the ears.
  * Maintain this position for 3 seconds.
  * Rest.
  * Repeat 10 times at the beginning of each hour during the immediate postoperative period on the hospital ward.
  * Suspend during the night.
  Arms: SHOULDER EXERCISES
Other: Hand exercises — Operational Definition:
  * Open and close the hands, making a fist and applying force.
  * Maintain this position for 3 seconds.
  * Rest.
  * Repeat 10 times at the beginning of each hour during the immediate postoperative period on the hospital ward.
  * Suspend during the night.
  Arms: HAND EXERCISES

SUMMARY:
This is a clinical trial aimed at understanding the impact of a shoulder exercise routine on postoperative shoulder pain in patients who have undergone laparoscopic hysterectomy.

**Main Questions:**

1. Does implementing a shoulder exercise routine immediately after laparoscopic hysterectomy reduce postoperative shoulder pain?

**Brief Explanation:** We want to see if doing shoulder exercises right after laparoscopic hysterectomy can help reduce the pain they might feel in their shoulders. This kind of pain can happen because of the gas used during the surgery. Using exercises could be a cost-effective and easy way to help patients recover better after the surgery.

**Hypothesis:** We think that doing shoulder exercises right after laparoscopic hysterectomy will lower the amount of shoulder pain patients experience after the surgery.

**Objective:** Our goal is to find out if a shoulder exercise routine can make a difference in how much shoulder pain patients have right after laparoscopic hysterectomy.

**How We'll Do It:** This study aims to evaluate the impact of a shoulder exercise routine on reducing postoperative shoulder pain in women who have undergone total laparoscopic hysterectomy at the National Institute of Perinatology. Recognizing the high prevalence and intensity of post-laparoscopy shoulder pain, the study compares the effectiveness of shoulder exercises to hand exercises in managing this pain. Patients, selected based on specific inclusion and exclusion criteria, will be randomly assigned to either the shoulder or hand exercise group. The exercise regimen involves performing specific movements at regular intervals during the immediate postoperative period, except at night. Pain intensity will be measured using a Visual Analog Scale at various intervals postoperatively. The study controls for several variables, including visceral and incisional pain, duration of pneumoperitoneum, analgesic use, and patient characteristics like BMI and comorbidities, to ensure a comprehensive understanding of the exercises' effectiveness. The hypothesis tests whether shoulder exercises can reduce shoulder pain more effectively than hand exercises. This research could have significant implications for enhancing recovery and pain management strategies post-laparoscopy.

DETAILED DESCRIPTION:
Main Objective

To evaluate the effect of a shoulder exercise routine versus a hand exercise routine on the intensity of shoulder pain in women postoperatively following total laparoscopic hysterectomy at the National Institute of Perinatology

Specific Objectives:

1. Describe the frequency and intensity of shoulder pain in women postoperatively following total laparoscopic hysterectomy.
2. Determine the effect of the shoulder exercise routine versus a hand exercise routine on the intensity of shoulder pain in women postoperatively following total laparoscopic hysterectomy.
3. Evaluate the adjusted effect of the proposed intervention on pain after identifying potential confounding variables. Postoperative management will be similar in both intervention groups, so we do not expect to make adjustments. In the event that confounding variables are identified, we will address them accordingly.

Hypothesis:

H0 (Null Hypothesis): Shoulder exercises in the postoperative period do not reduce shoulder pain by at least one point on the Visual Analog Scale compared to a hand exercise routine.

Description of the Procedure

Only patients scheduled for surgery at 8:00 AM will be considered to ensure that the exercise routine has a consistent duration for all patients during the postoperative period. Inclusion criteria involve patients receiving mixed anesthesia, and all patients will be positioned on the surgical table with shoulder pads and a hip angulation of 15 degrees with inflatable leg supports. Patients with negative pressure drains will be excluded from the study. The principal investigator will be blinded to the randomization group, and patient assessments will be conducted by another investigator.

Once a patient agrees to participate in the project and signs the informed consent authorization, they will be randomized into one of the treatment groups. Randomization will be done using opaque, sealed envelopes contained in a box. Each envelope will specify the assigned intervention group. An equal number of envelopes for both intervention groups will be prepared in advance and shuffled. Patients will choose an envelope. The box with envelopes will be safeguarded by the principal investigator using a simple randomization method generated by envelopes from an Excel-generated number table, distributed in sets of 8 until reaching the total of 112 patients.

Patients randomized to the exercise routine group will be instructed, upon recovery, about the exercise routine. The routine consists of lifting the shoulders as high as possible towards the ears, holding for 3 seconds, and then resting. This should be repeated 10 times at the beginning of each hour during the immediate postoperative period while on the hospital ward. The routine will be suspended during the night. The procedure will be standardized, as the principal investigator will personally explain and demonstrate it to all involved individuals who are responsible for explaining it to the patients. Telephone and in-person reminders will be made, and pain in the shoulders, incisions, and perineum will be recorded upon leaving the recovery room, at 6 hours and 24 hours postoperatively, as well as during the follow-up consultations on day 7 and day 30 post-surgery.

A data recording sheet with a visual analog scale from 0 to 10, representing the pain graphically, will be used to document pain levels upon leaving recovery, at 6 and 24 hours postoperatively, along with the time and dosage of analgesics and any rescue analgesics used. Additionally, patient adherence to the exercise routine will be recorded, allowing them to document their hospitalization days and the hours of the day when they perform the exercises.

Population: Patients postoperatively following uncomplicated total laparoscopic hysterectomy for benign conditions in the Department of Gynecology at INPer (National Institute of Perinatology).

Sample Type: Random consecutive cases, generated using a random number table in Excel.

Sample Size: Calculated using a formula for the difference in means of independent samples, considering a reported Visual Analog Scale (VAS) taing into account an VAS score reported at 6 hours postoperative witha mean in the experimental group of 3.0 (SD +-2.0) and the control group of 4.5 (SD +2.0) with a two tailed hypothesis, and statistical power 80% and an alphe error of 0.05% the sudy requiered a sample size of 28 per group plus 15% of possible dropout rate, the result is 33 patients per group and 66 in the total sample.

Sampling Type: Random consecutive cases.

Definition of Units of Observation: Patients postoperatively following uncomplicated total laparoscopic hysterectomy in the Department of Gynecology at INPer.

Definition of Control Group: Patients postoperatively following uncomplicated total laparoscopic hysterectomy in the Department of Gynecology at INPer, randomized to the control group, which will perform a series of hand exercises.

Inclusion Criteria:

- Patients undergoing uncomplicated total laparoscopic hysterectomy at INPer for benign pathology.

* Mixed anesthesia.
* Placement of shoulder pads on the surgical table during surgery.
* Adults who agree to participate and sign informed consent.

Exclusion Criteria:

* Patients with preoperative shoulder pain.
* Patients who had intraabdominal CO2 pressure greater than 15 mm Hg during surgery.
* Patients who received a postoperative analgesia pump.
* Patients participating in another protocol.

Elimination Criteria:

- Patients with postoperative complications requiring reoperation or Intensive Care Unit admission

x Dependent Variable:

Shoulder pain referred by the patient on a Visual Analog Scale (VAS) ranging from 0 to 10, at 6 hours, 24 hours, and 7 days postoperatively. The VAS is a tool used to help a person assess the intensity of certain sensations and feelings, such as pain. It consists of a straight line where one end represents the absence of pain, and the other end represents the worst imaginable pain. The patient marks a point on the line that corresponds to the amount of pain they feel in their shoulders.

Exercise Routine:

Two groups will be formed for the exercise routine:

1. Shoulder Exercises

   Operational Definition:

   - Lift the shoulders as high as possible toward the ears.

   - Maintain this position for 3 seconds.

   - Rest.

   - Repeat 10 times at the beginning of each hour during the immediate postoperative period on the hospital ward.
   * Suspend during the night.
2. Hand Exercises

Operational Definition:

* Open and close the hands, making a fist and applying force.
* Maintain this position for 3 seconds.
* Rest.
* Repeat 10 times at the beginning of each hour during the immediate postoperative period on the hospital ward.
* Suspend during the night.

Control Variables:

1. Visceral Pain Control

   Operational Definition:

   - Visceral pain (not at the surgical incision site) referred by the patient on a Visual Analog Scale (VAS) ranging from 0 to 10, at 6 hours, 24 hours, and 7 days postoperatively. The VAS is a tool used to help a person assess the intensity of certain sensations and feelings, such as pain. It consists of a straight line where one end represents the absence of pain, and the other end represents the worst imaginable pain. The patient marks a point on the line that corresponds to the amount of pain they feel.
2. Incisional Pain Control

Operational Definition:

* Pain at the surgical incision site referred by the patient on a Visual Analog Scale (VAS) ranging from 0 to 10, at 6 hours, 24 hours, and 7 days postoperatively. The VAS is a tool used to help a person assess the intensity of certain sensations and feelings, such as pain. It consists of a straight line where one end represents the absence of pain, and the other end represents the worst imaginable pain. The patient marks a point on the line that corresponds to the amount of pain they feel

Control Variables:

1. Duration of Neumoperitoneum

   Operational Definition:

   - Time in minutes of the duration of CO2 insufflation during the surgical event.
2. Average Neumoperitoneum Pressure

   Operational Definition:

   - Average pressure in millimeters of mercury (mm Hg) of CO2 used during the surgical procedure.
3. Use of Intravenous Analgesics in Immediate Postoperative Period

   Operational Definition:

   - Use of intravenous analgesics in the immediate postoperative period. This variable includes specific analgesics administered and their administration schedule.
4. Rescue Analgesic in Postoperative Period

   Operational Definition:

   - Use of an additional intravenous analgesic for uncontrolled pain in the immediate postoperative period.
5. Surgical Drainage

   Operational Definition:
   * Placement of any type of negative pressure drainage in the abdominal cavity.
6. Age

   Operational Definition:
   * The age of the patient in years.
7. Body Mass Index (BMI)

   Operational Definition:
   * BMI is a measure of the association between a person's weight and height, calculated as weight in kilograms divided by height in square meters.

   Control Variables (Continued):

12) Comorbidities

Operational Definition:

- Existence of a chronic disease in the patient at the time of surgery. This variable includes specific chronic diseases such as hypertension, diabetes, kidney disease, cardiovascular disease, psychiatric conditions, lung disease, immunosuppression, chronic pain syndrome, and other chronic diseases.

13) Chronic Pain Syndrome

Operational Definition:

- Presence of chronic pain that can range from mild to severe and persists or evolves for a long period of time (3 months or more).

14) Treatment with Psychotropic Drugs

Operational Definition:

- Use of medications for the treatment of mental illnesses or alterations of the psychic sphere.

15) Depression

Operational Definition:

- Assessed using a self-administered questionnaire with 14 items, divided into two subscales of seven items each: one for anxiety (odd-numbered items) and one for depression (even-numbered items). Responses are scored on a Likert scale ranging from 0 to 3, resulting in a minimum score of 0 and a maximum score of 21 for each subscale. Based on the scale, it is determined if the person has symptoms of anxiety or depression, to what extent, and whether it constitutes a clinical diagnosis. The scale is validated in Mexico.

16) Anxiety

Operational Definition:

- Assessed using the same questionnaire as for depression (15), with a Likert scale ranging from 0 to 3. The presence and level of anxiety symptoms are determined based on the scores.

17) Surgeon

Operational Definition:

- The gynecologist trained in gynecological endoscopic surgery who performs the total laparoscopic hysterectomy at the National Institute of Perinatology. The study includes various surgeons who perform these procedures.

18) Bleeding

Operational Definition:

- Blood loss during the surgical procedure, measured in milliliters (mL).

19) Adherence to Exercises

Operational Definition:

- Adherence to the exercise routine, measured as a percentage of exercises completed during the hospitalization.

T A) Independent Variable: Exercise Routine, Two Groups will be Formed

1. Shoulder Exercises Operational Definition: Lift the shoulders as high as possible towards the ears, hold for 3 seconds, and rest. Repeat 10 times at the beginning of each hour during the immediate postoperative period on the hospital floor. Suspend during the night.
2. Hand Exercises Operational Definition: Open and close the hands while making a fist, hold for 3 seconds, and rest. Repeat 10 times at the beginning of each hour during the immediate postoperative period on the hospital floor.

B) Dependent Variable: Shoulder Pain Reported by the Patient on a Visual Analog Scale (VAS) from 0 to 10, at 6 hours, 24 hours, and 7 days post-surgery.

* Type of Variable: Quantitative Continuous
* Measurement Level: 0-10

C) Control Variables: Bleeding, Surgeon, Anxiety, Depression, Treatment with Psychotropic Drugs, Chronic Pain Syndrome, Comorbidities, Body Mass Index, Age, Surgical Drainage, Rescue Analgesic Use, Standard Analgesic Regimen, CO2 Insufflation Pressure, Duration of Pneumoperitoneum

.

A) Independent Variable: Exercise Routine, Two Groups will be Formed

1. Shoulder Exercises Operational Definition: Lift the shoulders as high as possible towards the ears, hold for 3 seconds, and rest. Repeat 10 times at the beginning of each hour during the immediate postoperative period on the hospital floor. Suspend during the night.
2. Hand Exercises Operational Definition: Open and close the hands while making a fist, hold for 3 seconds, and rest. Repeat 10 times at the beginning of each hour during the immediate postoperative period on the hospital floor.

B) Dependent Variable: Shoulder Pain Reported by the Patient on a Visual Analog Scale (VAS) from 0 to 10, at 6 hours, 24 hours, and 7 days post-surgery.

* Type of Variable: Quantitative Continuous
* Measurement Level: 0-10

C) Control Variables: Bleeding, Surgeon, Anxiety, Depression, Treatment with Psychotropic Drugs, Chronic Pain Syndrome, Comorbidities, Body Mass Index, Age, Surgical Drainage, Rescue Analgesic Use, Standard Analgesic Regimen, CO2 Insufflation Pressure, Duration of Pneumoperitoneum

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing uncomplicated total laparoscopic hysterectomy at INPer for benign pathology.
* Mixed anesthesia.
* Placement of shoulder pads on the surgical table during surgery.
* Adults who agree to participate and sign informed consent.

Exclusion Criteria:

* Patients with preoperative shoulder pain.
* Patients who had intraabdominal CO2 pressure greater than 15 mm Hg during surgery.
* Patients who received a postoperative analgesia pump.
* Patients participating in another protocol

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Shoulder pain | 6 hours, 24 hours, and 7 days postoperatively
  Shoulder pain referred by the patient on a Visual Analog Scale (VAS) ranging from 0 to 10. The VAS is a tool used to help a person assess the intensity of certain sensations and feelings, such as pain. It consists of a straight line where one end represents the absence of pain, and the other end represents the worst imaginable pain. The patient marks a point on the line that corresponds to the amount of pain they feel in their shoulders.

SECONDARY OUTCOMES:
Visceral Pain | 6 hours, 24 hours, and 7 days postoperatively
  Visceral pain referred by the patient on a Visual Analog Scale (VAS) ranging from 0 to 10. The VAS is a tool used to help a person assess the intensity of certain sensations and feelings, such as pain. It consists of a straight line where one end represents the absence of pain, and the other end represents the worst imaginable pain. The patient marks a point on the line that corresponds to the amount of pain they feel in the abdomen (not in the incisions).
Incisional Pain | 6 hours, 24 hours, and 7 days postoperatively
  Incisional pain referred by the patient on a Visual Analog Scale (VAS) ranging from 0 to 10. The VAS is a tool used to help a person assess the intensity of certain sensations and feelings, such as pain. It consists of a straight line where one end represents the absence of pain, and the other end represents the worst imaginable pain. The patient marks a point on the line that corresponds to the amount of pain they feel in the incisions.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Perinatology, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Yang SC, Chang KY, Wei LF, Shyr YM, Ho CM. To drain or not to drain: the association between residual intraperitoneal gas and post-laparoscopic shoulder pain for laparoscopic cholecystectomy. Sci Rep. 2021 Jun 1;11(1):7447. doi: 10.1038/s41598-021-85714-4. PMID 34059697
- [Background] Lee DH, Song T, Kim KH, Lee KW. Incidence, natural course, and characteristics of postlaparoscopic shoulder pain. Surg Endosc. 2018 Jan;32(1):160-165. doi: 10.1007/s00464-017-5651-5. Epub 2017 Jun 22. PMID 28643053
- [Background] Wada S, Fukushi Y, Nishimura M, Matsumoto S, Takimoto K, Imai K, Ota H, Tsuzuki Y, Nakajima A, Fujino T. Analysis of risk factors of postlaparoscopic shoulder pain. J Obstet Gynaecol Res. 2020 Feb;46(2):310-313. doi: 10.1111/jog.14156. Epub 2020 Jan 20. PMID 31958892
- [Background] van Dijk J, Dedden SJ, Geomini P, van Kuijk S, van Hanegem N, Meijer P, Bongers MY. Randomised controlled trial to estimate reduction in pain after laparoscopic surgery when using a combination therapy of intraperitoneal normal saline and the pulmonary recruitment manoeuvre. BJOG. 2018 Oct;125(11):1469-1476. doi: 10.1111/1471-0528.15207. Epub 2018 Apr 15. PMID 29498786
- [Background] Reeve J, Stiller K, Nicol K, McPherson KM, Birch P, Gordon IR, Denehy L. A postoperative shoulder exercise program improves function and decreases pain following open thoracotomy: a randomised trial. J Physiother. 2010;56(4):245-52. doi: 10.1016/s1836-9553(10)70007-2. PMID 21091414
- [Background] Klein I, Kalichman L, Chen N, Susmallian S. A pilot study evaluating the effect of early physical therapy on pain and disabilities after breast cancer surgery: Prospective randomized control trail. Breast. 2021 Oct;59:286-293. doi: 10.1016/j.breast.2021.07.013. Epub 2021 Jul 21. PMID 34340163
- [Background] Tanner TN, Hall BR, Oran J. Pneumoperitoneum. Surg Clin North Am. 2018 Oct;98(5):915-932. doi: 10.1016/j.suc.2018.06.004. PMID 30243453
- [Background] Yamamoto-Furusho JK, Sarmiento-Aguilar A, Garcia-Alanis M, Gomez-Garcia LE, Toledo-Maurino J, Olivares-Guzman L, Fresan-Orellana A. Hospital Anxiety and Depression Scale (HADS): Validation in Mexican Patients with Inflammatory Bowel Disease. Gastroenterol Hepatol. 2018 Oct;41(8):477-482. doi: 10.1016/j.gastrohep.2018.05.009. Epub 2018 Jun 21. English, Spanish. PMID 29937084
- [Background] Bastamizad N, Abbasi P, Salari N, Jalali R. Comparing the Effect of Incentive Spirometry and Deep Breathing Exercises on the Level of Shoulder Pain and Nausea Following Laparoscopic Cholecystectomy Surgery: A Clinical Trial Study. Gastroenterol Nurs. 2023 Jan-Feb 01;46(1):14-22. doi: 10.1097/SGA.0000000000000720. Epub 2023 Jan 10. PMID 36706138
- [Background] Zeeni C, Chamsy D, Khalil A, Abu Musa A, Al Hassanieh M, Shebbo F, Nassif J. Effect of postoperative Trendelenburg position on shoulder pain after gynecological laparoscopic procedures: a randomized clinical trial. BMC Anesthesiol. 2020 Jan 29;20(1):27. doi: 10.1186/s12871-020-0946-9. PMID 31996139
- [Result] Choi JB, Kang K, Song MK, Seok S, Kim YH, Kim JE. Pain Characteristics after Total Laparoscopic Hysterectomy. Int J Med Sci. 2016 Jul 5;13(8):562-8. doi: 10.7150/ijms.15875. eCollection 2016. PMID 27499688